CLINICAL TRIAL: NCT05792657
Title: The ABEL Feasibility Study (Adherence, Better Health, Exercise and Life Satisfaction): A Randomized Controlled Trial
Brief Title: The ABEL Feasibility Study (Adherence, Better Health, Exercise and Life Satisfaction)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Norges idrettshøgskole (Other)
Collaborators: Kristiania University College (Other); ABEL Technologies (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: EMT2023
Record Dates: First submitted 2023-02-10; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-02

CONDITIONS: Obesity
Keywords: Exercise is medicine; Exercise adherence; Total physical activity level; Exercise professionals; Women with obesity (>30 BMI)
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Masking Description: Each participant will be randomly assigned (1:1:1:1) to one intervention group, HIGH, MEDIUM, LOW or CONTROL following a simple computer-based randomization program. All participants included in the study will conduct the baseline assessments before the randomization procedure. The study design will not allow for further masking of study participants or the exercise professional (caregivers to the interventions). Those from the research group involved in inclusion of the participants or follow-up measurements will not have access to the group allocation list. Further, all measurements will be completed and plotted without the research group information of group allocation. The statistical analyses will be done in SPSS, following a predefined analysis plan and before unmasking the study arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HIGH dosage in-person exercise coaching (Experimental): One in-person exercise session with an exercise professional/weekly. A total of 20 hours of in-person coaching during the 20 weeks of intervention.
  Interventions: Behavioral: High dosage in-person exercise coaching
- MEDIUM dosage in-person exercise coaching (Experimental): Two in-person exercise session with an exercise professional/monthly, and 15 minutes web-based behavioral support on the non-supervised weeks.A total of 10 hours in-person coaching during the 20 weeks intervention.
  Interventions: Behavioral: Medium dosage in-person exercise coaching.
- LOW dosage in-person exercise coaching (Experimental): One in-person exercise session with the exercise professional/monthly, and 15 minutes web-based behavioral support on the non-supervised weeks.Total of five hours of in-person coaching during the 20 weeks intervention.
  Interventions: Behavioral: Low dosage in-person exercise coaching
- CONTROL (No Intervention): Will be asked to continuing with normal life, and will receive regular follow-up care from their GP. This group will be giving the "Norwegian Directorate of Health's" recommendations for physical activity and nutrition, and will have access to the ABEL-app in order to register physical activity and exercise, but will not be provided any coaching during the 20 weeks.

INTERVENTIONS:
Behavioral: High dosage in-person exercise coaching — High dosage (one hour each week) of in-person exercise coaching by an exercise professional.
  Arms: HIGH dosage in-person exercise coaching
Behavioral: Medium dosage in-person exercise coaching. — Medium dosage (one hour every other week) of in-person exercise coaching by an exercise professional.
  Arms: MEDIUM dosage in-person exercise coaching
Behavioral: Low dosage in-person exercise coaching — Low dosage (one hour every month) of in-person exercise coaching by an exercise professional
  Arms: LOW dosage in-person exercise coaching

SUMMARY:
The ambition of the ABEL feasibility study is to test new "green prescription" follow-up models that can get more women with obesity, regularly active, with improved health and physical fitness. The project will evaluate the effect on exercise behavior, total physical activity level and mental and physical health outcomes by four different follow-up models by an exercise professional: HIGH-dosage in-person exercise coaching (four session monthly), MEDIUM- dosage in-person exercise coaching (two sessions monthly) LOW-dosage in-person exercise coaching (one session monthly). The main aim of this study is to evaluate which of these follow-up models is most effective on improving women's exercise adherence, total physical activity level, physical fitness, and mental and physical health. This will be weighed against the cost of each of the follow-up models, in order to identify the best model from a socioeconomic cost-effectiveness perspective. Moreover, the study will identify potential barriers among patients, General Practitioners and exercise professionals that prevents optimal outcome from the current green prescription model.

DETAILED DESCRIPTION:
BACKGROUND:

Obesity, defined as "abnormal or excessive fat accumulation that presents a risk to health" and a body mass index (BMI) of ≥30, represents a major health challenge and economic burden for welfare systems worldwide. Living with obesity is reported to account for 80-85% of the risk of developing non-communicable diseases such as diabetes type 2. Guidance on regular physical activity, exercise and healthy eating is traditionally the first measure taken for patient who undergo treatment for obesity. Treatment for obesity in the primary healthcare service is largely coordinated by general practitioners (GP). Green prescriptions (tailored advice and guidance on lifestyle factors related to development of disease, such as physical activity and healthy eating) can be prescribed as a treatment alternative to patients with chronic disease, such as obesity. However, few GPs in Norway use green prescriptions as a treatment alternative to their patients, and 41% of GPs in 2006 reported that they had newer prescribed green prescriptions to their patients. The lack of sufficient follow-up of patients has been reported as a main limitation with the current green prescription model.

Previous research underlines the importance in-person coaching for patients who receives green prescriptions, as well as establishing collaborations with professions such as exercise professionals to be able to provide sufficient coaching of patients. Hence, in-person coaching by an exercise professional may have the means to get more patients with obesity regularly active, and can potentially be the follow-up alternative the current green prescription model is lacking.

However, considering the expenses and practical considerations associated with in-person coaching, has former studies displayed the advantage of using web-based behavioral support for patients with obesity. Yet, web-based behavioral support often proves to have poor completion rate, and need to be combined with face-to-face guidance and feedback in order to increase adherence. However, when combining in-person coaching and web-based behavioral support, there is still limited knowledge on how frequent in-person coaching needs to occur, in order to increase adherence. More knowledge on frequency of follow-up is essential for an approach towards an economical sustainable green prescription model.

AIMS:

1. In women with obesity (BMI≥30), what is the effect of in-person exercise coaching (high vs. medium vs. low dosage) on exercise adherence and total physical activity level?
2. In women with obesity (BMI≥30), what is the effect of in-person exercise coaching (high vs. medium vs. low dosage) on mental health variables (quality of life, self-efficacy and barriers and motivation to exercise)?
3. In women with obesity (BMI≥30), what is the effect of in-person exercise coaching (high vs. medium vs. low dosage) on health (glycated hemoglobin, cholesterol, blood pressure, waist circumference, BMI and urinary incontinence) and physical fitness (aerobic endurance, muscular strength)?
4. Is adherence to exercise and succeeding health effects associated with the exercise professionals level of education and knowledge base?
5. What are the participant's experiences, barriers and facilitators of participating in the ABEL-project?
6. What are the general practitioners' experiences, barriers and facilitators of using the "green prescription"?

STUDY DESIGN AND METHOD:

In the present feasibility study, women with obesity (BMI of ≥30, n=200) will be recruited to a 20-week randomized control trial (RCT) with four arms. Participants will be recruited via social media platforms (Facebook and Instagram). Using simple computer-based randomization program, participants will be randomized to one of the following arms: HIGH dosage in person exercise coaching, MEDIUM dosage in-person exercise coaching, LOW dosage in-person exercise coaching, and CONTROL group. A total of 25 exercise professionals, working full time as a personal trainer will follow up the participants at one of the following fitness clubs: "Feel24", "PT-group", "Nr1 Fitness", "Trento" or "Spenst". All participants in the intervention arms (HIGH, MEDIUM and LOW) groups are provided the same frequency (each week) of follow-up by the exercise professional. At baseline, all participants will respond to an electronic questionnaire, perform measures of muscular strength and aerobic endurance, measure blood pressure, hip-waist ratio, BMI (height and weight) and take a blood sample (Tigeni Kit). After a 20-weeks intervention period, participants will perform a post-test including the same previous mentioned outcome measures.

n=15 of women from intervention arms HIGH (n=5), MEDIUM (n=5) and LOW (n=5), will also be invited to participate in an in-depth interview in order to investigate participants experiences and barriers for participating in the ABEL feasibility study.

In addition to the RCT, the project will also recruit GPs (n=8) to participate in an in-depth interview with researchers from the project group. GPs will be recruited to provide more in-depth understanding on reasons for what the current green prescription model is lacking.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 65 years
* No fitness club membership six months prior to recruitment
* Low-active (<150 minutes of moderate-intensity or 75 minutes of vigorous-intensity per week)
* Norwegian speaking
* In possession of a mobile phone.

Exclusion Criteria:

* Chronic disease or pathology (e.g severe hypertension 180/110 mm Hg), heart disease or lung disease hindering exercise
* Changing GP during the intervention
* Functional impairment due to injuries hindering physical activity and exercise.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2023-06-26 (Estimated); Study Completion 2023-06-26 (Estimated)

PRIMARY OUTCOMES:
Adherence (attendance) to prescribed exercise sessions | Continuously during the intervention period of 20 weeks
  Measures of adherence to exercise sessions will be collected through the ABEL-app (ABEL Technologies). Sessions performed with the exercise professional will be logged through the ABEL-app of the exercise professional, while sessions performed independently will be logged through the ABEL-app of the participant. Participants adherence will be measured by attendance (percentage of exercise sessions completed out of exercise sessions offered).

SECONDARY OUTCOMES:
Fulfillment of physical activity recommendations | At baseline and following the intervention period (20 weeks)
  To determine whether participants are meeting the physical activity recommendations, a single question whil be asked : "for the last six months, have you participated in more or less than 150 minutes of moderate physical activity each week?" Participants can respond either "more" or "less", where more is greater than less. Fulfillment of physical activity recommendations, exercise frequency, duration of exercise sessions and physical activity mode will be combined in order to measure participants physical activity behavior.
Exercise frequency | At baseline and following the intervention (20 weeks).
  Exercise frequency will be measured by a single questions: "how often do you exercise each week?" participants can give a respond from 0-"7, where 7 is greater than 0. Exercise frequency, fulfillment of physical activity recommendations, duration of exercise sessions and mode of physical activity will be combined in order to measure participants physical activity behavior.
Duration of exercise sessions | At baseline and following the intervention period (20 weeks)
  Duration of exercise sessions will be measured by a single question: "how long do you usually exercise per session? Participants can give a respond in minutes from "below 30 minutes" to "above 90 minutes", where above 90 minutes is greater than 30 minutes. Duration of exercise sessions, fulfillment of physical activity recommendations, mode of physical activity and frequency of exercise sessions will be combined in order to measure participants physical activity behavior.
Mode of physical activity | At baseline and following the intervention period (20 weeks)
  To determine which type of physical activity participants performs, participants will answer a single question: "Which of the following types of activities do you usually participate in? Participants are able to select more than one response of: "Commuting activities", "activities at home", "cycling", "walking", "exercising at a fitness club", "home exercises", and "exercising in sports". Mode of physical activity, fulfillment of physical activity recommendations, exercise frequency and exercise durations will be combined to measure participants physical activity behavior.
Health-related quality of life | At baseline and following the intervention period (20 weeks)
  Will be measured by a Norwegian version of "The MOS 36-item short-form health survey" (SF-36). The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0-100. Lower scores = more disability, higher scores = less disability.
Self-efficacy | at baseline and following the intervention period (20 weeks)
  Will be measured by a Norwegian abbreviated validated version of a "Self-Efficacy Survey" consisting of 12 statements. The subscale covers four to eight statements where the participants rated each statement on a five-point scale, where 5 is the highest grade of self-efficacy, and 1 is the lowest. For each subscale, a sum score (from 1 to 5) will be calculated by adding scores from each statement, divided by the number of statements.
Motivation for exercise and physical activity | At baseline and following the intervention period (20 weeks)
  Will be measured by a Norwegian version of the validated survey "BREQ-2", which measures the levels of self-determination in motivation for exercise and physical activity on a 5-point Likert-scale (from 1 to 5). Score range from 0-100, where high scores means more intrinsic motivated for exercise and physical activity.
Perceived social support from family and friends | At baseline and following the intervention period (20 weeks)
  Questions to measure social support for exercise and physical activity will be based on a validated social support questionnaire consisting of 13 statements concerning social support from friends and family. The participants rate each statement on how often, on a five-point scale, their family or friends have been supportive of them exercising. A total social support score will be calculated (from 6 to 30), where higher scores demonstrated greater social support for exercise and physical activity.
Stage of motivational readiness for exercise and physical activity | At baseline and following the intervention period (20 weeks)
  Will be measured in line with a previously conducted questionnaire on exercise professionals effect on changing attitude towards physical activity and exercise. Participants will rate one statement (on how likely they are to start exercising the next six months) according to the five stages in the stages of change model: re-contemplation (not intending to make changes), Contemplation (considering a change), Preparation (getting ready to make a change), Action (actively engaged in making a change but only for a short while) & Maintenance (sustaining the change over time). "Maintenance" is the highest grade of motivation, followed by "Action", "Preparation" and "Contemplation". "Re-contemplation" is the lowest grade of motivation.
Barriers to exercise | At baseline and following the intervention period (20 weeks)
  Questions will be based on barriers previously identified among a Norwegian adult population (n= 12 504) and among fitness club members. 18 barriers will be included in the questionary. The participants rated how limiting they perceived each barrier to be on a three-point scale (1= not correct, 3=very correct). By adding the score from each barrier divided by the number of statements, a sum-score (from 1 to 3) for each subscale will be calculated.
Urinary incontinence | At baseline and following the intervention period (20 weeks)
  Will be measured using a Norwegian version of the "Incontinence Questionaire-Short Form (ICIQ-UI SF)". Measures will be given by a Likert scale from "never" to "all the time". Awareness and knowledge about pelvis floor muscles exercises will be assessed by single questions: "Do you do pelvic floor muscle exercises?" If yes, how many times weekly?" "If yes, has your exercise professional provided you any coaching on pelvic floor muscle exercises?"
Glycated hemoglobin | At baseline and following the intervention period (20 weeks)
  Will be collected through capillary blood drawn from finger pricks by Tigeni self testing kits. Measures will be given in mmol/L
Blood pressure | At baseline and following the intervention period (20 weeks)
  Will be assessed by the participants GP. Both systolic and diastolic blood pressure will be measured. Unit of measures is millimeters of mercury (mmHg).
Weight | At baseline and following the intervention period (20 weeks)
  Will be measured by the participants GP. Unit of measures is in kilogram (kg). Weight and height will be combined to report BMI in kg/m2
Height | At baseline and following the intervention period (20 weeks)
  Will be measured by the participants GP. Unit of measures is centimeters (cm). Weight and height will be combined to report BMI in kg/m2
Cholesterol | At baseline and following the intervention period (20 weeks)
  Cholesterol will be collected through capillary blood drawn from finger pricks by Tigeni self testing kits. Unit of measures is mmol/L
Heart rate recovery | At baseline and following the intervention period (20 weeks)
  Unit of measures is beats per minute (BPM). Heart rate recovery combined with RPE and working heart rate will be used to assess relative changes in participants aerobic endurance.
The Borg Rating of Perceived Exertion (RPE) | At baseline and following the intervention period (20 weeks)
  Measures will be given on a rating scale from 6 (no exertion) to 20 (maximal exertion). Participants will perform a standardized incline treadmill-walking test. RPE, heart rate recovery and changes in working heart rate will be combined to assess participants relative changes in aerobic endurance.
Working heart rate | At baseline and following the intervention period (20 weeks)
  Unit of measures is beats per minute (BPM). Working heart rate is combined with RPE and Heart rate recovery to assess participants relative changes in aerobic endurance.
Muscular strength | At baseline and following the intervention period (20 weeks)
  Will be assessed by a 1-RM (repetition maximum) estimation test in: chest press, close grip lat pull down and leg press. Load will progressively be increase until the participant reaches nine or less repetitions. Brzycki 1-RM prediction equation will be used to estimate the 1-RM based on the resistance and repetitions performed. The equation is mathematically expressed as 1RM = W/ [102.78- 2.78(R)]/100, where W is the weight used and R is the maximal number of repetitions performed.
Factors associated with exercise adherence and drop-out | Following the intervention period (20 weeks)
  n=15 of participants from the intervention group: HIGH, MEDIUM and LOW will be invited to participate in a semi-structured in-depth interview. A former investigation in Norway, including 14 questions designed to address factors associated with exercise adherence and drop-out. These questions will be combined with questions covering BPNES in order to measure participant's experiences, barriers and facilitators of participating in the study.
Basic physicological needs in exercise (BPNES) | Following the intervention period (20 weeks)
  n=15 of participants from the intervention group: HIGH, MEDIUM and LOW. Will be invited to participate in a semi-structured in-depth interview including questions covering fulfillment of BPNES (autonomy, relatedness and competence). Questions regarding fulfilment of BPNES will be combined with questions designed to address factors associated with exercise adherence and drop-out, to evaluate participant's experiences, barriers and facilitators of participating in the study.
In-depth interview (general practitioners) | Following the intervention period (20 weeks)
  n=8 general practitioners will participate in a semi-structured in-depth interview (approximately 45 min). The interview will be led by researchers from the project group, audiotaped and transcribed verbatim. Questions will be based on a previous qualitative study conducted on GPs in Norway, covering GPs experiences with the current green prescription model, and views on exercise as medicine.

CONTACTS AND LOCATIONS:
Overall Officials: Tron Krosshaug, PhD, Study Chair — Norwegian School of Sport Sciences
Locations (1):
- Norwegian School of Sport Sciences, Oslo, Norway

REFERENCES:
- [Background] O'Regan A, Pollock M, D'Sa S, Niranjan V. ABC of prescribing exercise as medicine: a narrative review of the experiences of general practitioners and patients. BMJ Open Sport Exerc Med. 2021 Jun 2;7(2):e001050. doi: 10.1136/bmjsem-2021-001050. eCollection 2021. PMID 34150320
- [Background] Elley CR, Garrett S, Rose SB, O'Dea D, Lawton BA, Moyes SA, Dowell AC. Cost-effectiveness of exercise on prescription with telephone support among women in general practice over 2 years. Br J Sports Med. 2011 Dec;45(15):1223-9. doi: 10.1136/bjsm.2010.072439. Epub 2010 Nov 16. PMID 21081641
- [Background] Ries AL, Kaplan RM, Myers R, Prewitt LM. Maintenance after pulmonary rehabilitation in chronic lung disease: a randomized trial. Am J Respir Crit Care Med. 2003 Mar 15;167(6):880-8. doi: 10.1164/rccm.200204-318OC. Epub 2002 Dec 27. PMID 12505859
- [Background] Powell-Wiley TM, Poirier P, Burke LE, Despres JP, Gordon-Larsen P, Lavie CJ, Lear SA, Ndumele CE, Neeland IJ, Sanders P, St-Onge MP; American Heart Association Council on Lifestyle and Cardiometabolic Health; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology; Council on Epidemiology and Prevention; and Stroke Council. Obesity and Cardiovascular Disease: A Scientific Statement From the American Heart Association. Circulation. 2021 May 25;143(21):e984-e1010. doi: 10.1161/CIR.0000000000000973. Epub 2021 Apr 22. PMID 33882682
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Gjestvang C, Abrahamsen F, Stensrud T, Haakstad LAH. Motives and barriers to initiation and sustained exercise adherence in a fitness club setting-A one-year follow-up study. Scand J Med Sci Sports. 2020 Sep;30(9):1796-1805. doi: 10.1111/sms.13736. Epub 2020 Jun 15. PMID 32488898
- [Background] Sallis JF, Grossman RM, Pinski RB, Patterson TL, Nader PR. The development of scales to measure social support for diet and exercise behaviors. Prev Med. 1987 Nov;16(6):825-36. doi: 10.1016/0091-7435(87)90022-3. PMID 3432232
- [Background] McClaran SR. The effectiveness of personal training on changing attitudes towards physical activity. J Sports Sci Med. 2003 Mar 1;2(1):10-4. eCollection 2003 Mar. PMID 24616604
- [Background] Sorensen M, Gill DL. Perceived barriers to physical activity across Norwegian adult age groups, gender and stages of change. Scand J Med Sci Sports. 2008 Oct;18(5):651-63. doi: 10.1111/j.1600-0838.2007.00686.x. Epub 2007 Dec 11. PMID 18086263
- [Background] Murcia JA, Gimeno EC, Camacho AM. Measuring self-determination motivation in a physical fitness setting: validation of the Behavioral Regulation in Exercise Questionnaire-2 (BREQ-2) in a Spanish sample. J Sports Med Phys Fitness. 2007 Sep;47(3):366-74. PMID 17641607
- [Background] Gron Jensen LC, Boie S, Axelsen S. International consultation on incontinence questionnaire - Urinary incontinence short form ICIQ-UI SF: Validation of its use in a Danish speaking population of municipal employees. PLoS One. 2022 Apr 6;17(4):e0266479. doi: 10.1371/journal.pone.0266479. eCollection 2022. PMID 35385519
- [Background] Moutao JM, Serra LF, Alves JA, Leitao JC, Vlachopoulos SP. Validation of the Basic Psychological Needs in Exercise Scale in a Portuguese sample. Span J Psychol. 2012 Mar;15(1):399-409. doi: 10.5209/rev_sjop.2012.v15.n1.37346. PMID 22379729
- [Background] Bringedal B, Aasland OG. [Doctors' use and assessment of a fee-for-service life-style advice scheme]. Tidsskr Nor Laegeforen. 2006 Apr 6;126(8):1036-8. Norwegian. PMID 16619061
- [Background] Brzycki M. Strength testing-predicting a one-rep max from reps-to-fatigue. Journal of Physical Education, Recreation & Dance. 1993;64(1):88-90.
- [Derived] Gjestvang C, Kalhovde JM, Mauseth Tangen E, Clemm H, Haakstad LAH. Impact of In-Person and Mobile Exercise Coaching on Psychosocial Factors Affecting Exercise Adherence in Inactive Women With Obesity: 20-Week Randomized Controlled Trial. J Med Internet Res. 2025 Feb 25;27:e68462. doi: 10.2196/68462. PMID 39999434

DOCUMENTS (1):
  • Study Protocol (2023-03-19): https://cdn.clinicaltrials.gov/large-docs/57/NCT05792657/Prot_000.pdf